CLINICAL TRIAL: NCT00589199
Title: Functional Electrical Stimulation for Production of Artificial Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Anthony F. Dimarco, Professor of Medicine, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB93-00133
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries; Paralysis
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Functional Electrical Stimulation for Production of Artificial Cough
  Interventions: Procedure: Placement and use of the device

INTERVENTIONS:
Procedure: Placement and use of the device — Surface electrodes currently used for peripheral muscle stimulation by other groups will be applied to the abdominal wall and over the posterior lower thoracic rib cage. Between two and three pairs (anodic and cathodic) of electrodes will be used in combination to activate the expiratory muscles. Electrodes will be positioned at various points over the abdominal wall and the posterior thoracic rib cage to ascertain optimal placement for airway pressure and expiratory airflow generation. The electrical stimulators to be used (EMPI and NeuroMedic) are powered by 9-volt batteries. These stimulators are currently in clinical use to stimulate other skeletal muscles and are known to be quite safe.

SUMMARY:
The purpose of the present study is to assess the utility of abdominal muscle stimulation to provide large positive airway pressures and expiratory airflow thus simulating cough. Restoration of cough in spinal cord injured patients may reduce the incidence of respiratory complications such as atelectasis, respiratory tract infections and respiratory failure.

DETAILED DESCRIPTION:
Cough is a complex defensive respiratory reflex mechanism necessary for the clearance of respiratory secretions and foreign materials. In patients with chronic bronchitis, previous investigations have found that the cough mechanism is the most effective measure to enhance mucous clearance from the lung.

Patients with cervical and thoracic spinal cord injuries have suffered a loss of the major portion of their expiratory muscles. Consequently, they are unable to generate significant positive intrathoracic airway pressures or airflow and have a markedly increased risk of developing pulmonary infections. Mechanical methods have been developed to enhance cough production. However, these have resulted in only marginal increases in airway pressure.

Preliminary studies in our laboratory in animal experiments and those of others in humans have suggested that the abdominal muscles can be stimulated directly by surface electrodes. The purpose of the present study, therefore, is to assess the utility of abdominal muscle stimulation in quadriplegics and paraplegics to simulate cough. A range of stimulus parameters and electrode locations will be assessed to determine optimal stimulus paradigms. Airway pressure and expiratory airflow will be used as indices of cough effectiveness. If successful, abdominal muscle stimulation may be a useful tool to restore cough and hopefully reduce the incidence of respiratory complications such as atelectasis and infection in spinal cord injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical or thoracic spinal cord injury

Exclusion Criteria:

* Significant cardiovascular disease
* Active lung disease
* Pacemaker or other metallic implant
* Legally incompetent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1993-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Measurements of airway pressure and expiratory flow rate to evaluate efficacy of cough | one year

SECONDARY OUTCOMES:
Incidence of respiratory complications | one year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F DiMarco, MD, Principal Investigator — MetroHealth Medical Center and Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States